CLINICAL TRIAL: NCT03634514
Title: National, Monocentric, Randomized, Double-blind, Controlled, Crossover Clinical Trial, to Evaluate the Non-inferiority of Pain Intensity After the Application of Recombinant Human Somatropin - Biomatrop (Biosintética Farmacêutica) in Relation to Recombinant Human Somatotropin - Hormotrop (Bergamo), Single Dose, in Healthy Subjects of Both Genders
Brief Title: Non-inferiority Evaluation of Pain Intensity After Biomatrop (Somatropin) Application in Relation to Hormotrop (Somatropin), in Healthy Subjects
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ache Laboratorios Farmaceuticos S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: PPES 002/18
Record Dates: First submitted 2018-08-13; First posted 2018-08-16 (Actual); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Application of Biomatrop (Experimental): A single dose of Recombinant Human Somatropin - Biomatrop is administered. The pain intensity is evaluated using visual analogue scale (0-10cm) and record the incidence of adverse events.
  Interventions: Drug: Recombinant human growth hormone - Biomatrop; Drug: Recombinant human growth hormone - Hormotrop
- Application of Hormotrop (Active Comparator): A single dose of Recombinant Human Somatropin - Hormotrop is administered. The pain intensity is evaluated using visual analogue scale (0-10cm) and record the incidence of adverse events.
  Interventions: Drug: Recombinant human growth hormone - Biomatrop; Drug: Recombinant human growth hormone - Hormotrop

INTERVENTIONS:
Drug: Recombinant human growth hormone - Biomatrop — The subjects who recieve Biomatrop first, after a period maximum of 24 hours will recieve a dose of Hormotrop.
Drug: Recombinant human growth hormone - Hormotrop — The subjects who recieve Hormotrop first, after a period maximum of 24 hours will recieve a dose of Biomatrop.

SUMMARY:
Randomized, Double-blind, Controlled, Crossover, in which 68 subjects (34 males and 34 females) will receive, in each stage, an application of 4 UI, subcutaneous, single dose, of the investigational drug (Recombinant Human Somatropin - Biomatrop) and the comparator (Recombinant Human Somatropin - Hormotrop) according to randomization to evaluate the Non-inferiority of Pain Intensity After the Application of Hormotrop, using Visual Analogue Scale (0-10cm) and record the incidence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Skin phototype from 2 to 4, according to Fitspatrick classification: http://www.sbd.org.br/dermatologia/pele/cuidados/classifica cao-dos-fototipos-de-pele/ ;
* Subjects with normal laboratory, type 1 urine exam, vital signs and ECG results;
* Weight ≥ 50kg and Body Mass Index ≤ 30 ;
* Healthy subject according with clinical history
* Ability to understand and consent their participation in this clinical study, expressed by signing the Informed Consent Form (ICF);
* Subject who have negative results for stool protoparasitological examination accomplished in clinical study. Subjects with positive results for Endolimax nana, Entamoeba hartmanni, Entamoeba coli, Iodamoeva btshlii, Chilomastix mesili, Trichomonas hominis, Retortamonas intestinalis e Enteromonas hominis will be able to be included in the study. At the end of the study those subjects will be guided to treatment according to clinic investigator criteria.

Exclusion Criteria:

* Laboratory and clinical exam results out of normal range values, unless considered by physician clinically irrelevant;
* Positive sorology for HIV;
* Positive sorology for Hepatitis B;
* Positive sorology for Hepatitis C;
* Known hypersensitivity to the components of the medicines used during the study or related chemical compounds;
* Subjects that has participated in clinical trial protocols in the last twelve (12) months (National Board of Health- Resolution 251 of 07 August 1997, Part III, sub-item J), unless the investigator considers that there may be a direct benefit to it;
* Use of any type of regular medication within two (2) weeks or five (5) half-lives (whichever lasts longer) before administration of the first dose of the investigational product (IP). The eventual use of medication, which in the opinion of the Principal Investigator or physician does not interfere with the pharmacokinetics of IP in study will not be considered as exclusion criteria;
* History of alcohol abuse or having ingested alcoholic drink 24 hours prior to IP administration;
* History of psychotropic drug use and / or positive outcome for any of the components of the drug abuse test for amphetamine, benzoylecgonine (cocaine), benzodiazepines, methamphetamine, opiates, morphine, etrahydrocannabinol-THC (Marijuana / Marijuana). Subjects who used marijuana and hashish in less than three months before the consultation will be excluded. For drugs like cocaine, crack and heroin will be excluded subjects who present any use history;
* Any finding of clinical observation, laboratory abnormality or therapy which, in the opinion of the investigator, may put the subject at risk or interfere with the purpose of the study;
* The subject have any condition that in investigator's opinion prevents him/her from participating in the study;
* History of food allergy or hyperactivity to medications or food;
* Regular smokers or ex-smokers who have stopped for less than 6 months;
* Subjects who have a relationship of kinship to second degree or any bond with the sponsor or research center employees;
* Subjects with the following ECG changes: sinus tachycardia with heart rate ˃ 120 bpm; bradycardia sinus heart rate <50 bpm; atrial tachycardia, ventricular or junctional; ectopic atrial rhythm; atrial fibrillation; atrial flutter; accelerated idioventricular rhythm; locking atrium ventricular (BAV) of 1º, 2º and 3º degrees; ventricular pre-excitation; complete blockage of right or left branch; rhythm of pacemaker; supraventricular tachycardia (nodal tachycardia, ventricular atrial tachycardia) or any other clinically significant;
* Male subjects who do not agree to use acceptable contraceptive methods: (a) contraceptive methods for the participant: barrier preservative, except for (vasectomy) or for participants who declare that they do not engage in sexual practices or exercise them non-reprodutively; (b) contraceptive methods for the partner: oral contraceptive, intravenous contraceptive, intrauterine device (IUD), hormonal implant, hormonal transdermal patch, tubal ligation, and barrier methods except for female partners that are surgically sterile (bilateral oophorectomy or hysterectomy), or menopause for at least 01 (one) year;
* Women who do not agree to use acceptable contraceptive methods (oral contraceptive, intravenous contraceptive, intrauterine device (IUD), hormonal implant, barrier methods, hormonal transdermal patch and tubal ligation); except for those surgically sterile (bilateral oophorectomy or hysterectomy), menopause for at least one year, and participants who report not engaging in sexual practices or non-reproductive practices;
* Women in pregnancy or nursing period.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Estimated)
Dates: Start 2018-08-27 (Estimated); Primary Completion 2018-09 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | 1 hour
  Report the Pain Intensity using Visual Analogue Scale (0-10cm)

CONTACTS AND LOCATIONS:
Overall Officials: Sérgio Alberto Cunha Vêncio, Principal Investigator — Instituto de Ciências Farmacêuticas (ICF)
Locations (1):
- Instituto de Ciências Farmacêuticas, Goiânia, Goiás, Brazil